CLINICAL TRIAL: NCT06392412
Title: Effects of Fully Immersive Virtual Reality Cognitive Training Based on Instrumental Activities of Daily Living for Older Adults With Mild Cognitive Impairment
Brief Title: Virtual Reality Cognitive Training for Older Adults With Mild Cognitive Impairment
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Da-Yeh University (Other)
Responsible Party: Principal Investigator, I-Chen Chen, Assistant Professor, Da-Yeh University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DaYehU
Record Dates: First submitted 2024-04-26; First posted 2024-04-30 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Mild Cognitive Impairment; Older Adults
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR Group (Experimental)
  Interventions: Behavioral: fi-VR Cognitive Training
- Control Group (Active Comparator)
  Interventions: Behavioral: Traditional Cognitive Training

INTERVENTIONS:
Behavioral: fi-VR Cognitive Training — All participants will 16 sessions over eight weeks, with two sessions per week, each lasting 70 minutes. Participants in the fi-VRCT will use the virtual reality system with head-mounted display and handheld controllers. The fi-VRCT will be administered by an experienced research assistant.
  Arms: VR Group
Behavioral: Traditional Cognitive Training — All participants will 16 sessions over eight weeks, with two sessions per week, each lasting 70 minutes. The CT control program will include cognitive board games designed to improve various cognitive capacities. Certified community occupational therapists will lead the CT control group.
  Arms: Control Group

SUMMARY:
This study aims to (1) develop and assess the feasibility of a fi-VRCT program based on IADL for older adults with MCI, (2) implement and evaluate the effectiveness of the fi-VRCT program based on IADL in older adults with MCI, and (3) investigate the potential mechanism of the fi-VRCT program based on IADL for older adults with MCI and refine this intervention accordingly.

DETAILED DESCRIPTION:
As research on cognitive training methods for older adults with mild cognitive impairment (MCI) progresses, fully immersive virtual reality cognitive training (fi-VRCT) has emerged as a promising approach. While the benefits of fi-VRCT for enhancing cognitive function have been recognized, its potential to improve instrumental activities of daily living (IADL) and promote independence remains uncertain. This study addresses these questions by developing and validating a fi-VRCT program based on IADL to enhance cognitive and IADL performance among older adults with MCI.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 65 or above.
2. MoCA score between 18 and 25.
3. Capability to follow directions and do tasks.

Exclusion Criteria:

1. History of dementia.
2. Previous neurodegenerative illness diagnosis.
3. Severe medical or surgical problems.
4. Major psychological disorders.
5. Inability to use VR system

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes scores of Montreal Cognitive Assessment (MoCA) | At baseline, at week 9, and at 3-month follow-up.
  The MoCA comprises12 items, it assesses orientation to time and place, attention, concentration, short-term memory, \working memory, visuospatial abilities, language, and executive function. Scores on the MoCA range from 0 to 30, with a higher score indicative of better global cognition. A total score of 26 or above is considered within the normal cognitive function range, while a total score of 18 to 25 indicates mild cognitive impairment
Change scores of Wechsler Memory Scale (WMS) | At baseline, at week 9, and at 3-month follow-up.
  The Wechsler Memory Scale is a neuropsychological test designed to assess memory in adults aged 16 to 90. Family Pictures, Spatial Span, and Word List will be used to evaluate visual, auditory, immediate, delayed, and working memory. For each subtest, higher scores indicate better performance in memory performance. Based on age ranges, raw scores will be transformed into scaled scores ranging from 1 to 19.
Change scores of Amsterdam Instrumental Activities of Daily Living Questionnaire, Short Version | At baseline, at week 9, and at 3-month follow-up.
  The questionnaire is informant-reported and is typically completed by a caregiver. It comprises 30 items in seven categories: household activities, household appliances, finances, work, computer use, appliances, and leisure activities. Each item is rated based on the difficulty levels in performing it, ranging from no difficulty in performing the task to no longer being able to perform it. Score ranges from 0 to 100 and lower score indicates better functional ability.
Change scores of Lawton Instrumental Activities of Daily Living | At baseline, at week 9, and at 3-month follow-up.
  The Lawton Instrumental Activities of Daily Living is commonly employed to assess participants' ability to perform daily tasks and identify early functional decline. In semi-structured interviews, participants describe how they currently perform the eight IADLs. Each item is rated based on the levels of competence, ranging from independence in performing the activity to not being able to perform it at all. Score ranges from 8 to 31 and higher scores indicate better functional ability.

SECONDARY OUTCOMES:
Change scores of Digit Span | At baseline, at week 9, and at 3-month follow-up.
  Participants will be verbally presented with a random series of digits and asked to repeat them in the same order presented (forward span), in the reverse order (backward span), or ascending order (serial span). The raw score is determined by the number of the correct items and is transformed into a scaled score ranging from 1 to 19. Higher scores indicate better performance.
Change scores of Stroop Color-Word Test | At baseline, at week 9, and at 3-month follow-up.
  The examinee is instructed to read words or to name the ink colors as quickly as possible within a specified time limit. The Stroop Color-Word Test consists of congruent and incongruent stimuli. Reaction time and errors on congruent and incongruent trials are recorded. A more minor time difference between congruent and incongruent trials indicates better executive function

OTHER OUTCOMES:
Presence Questionnaire | The initial, second, fifth, ninth, thirteenth, and final intervention sessions.
  The questionnaire evaluates the extent to which participants feel a sense of presence within the virtual environment. It comprises 17 items grouped into three categories: involved/control, natural, and interface quality. It employs a seven-point Likert scale, and the score ranges from 17 to 119. Higher scores indicate a stronger sense of presence.
Immersive Tendencies Questionnaire | The initial, second, fifth, ninth, thirteenth, and final intervention sessions.
  The questionnaire measures participants' capacity to immerse or engage in the virtual environment fully. It comprises 16 items distributed across three subscales: involvement, focus, and games. It employs a seven-point Likert scale, the score ranges from 16 to 112. Higher scores indicate a greater tendency to become immersed.
Simulator Sickness Questionnaire | The initial, second, fifth, ninth, thirteenth, and final intervention sessions.
  The questionnaire assesses any adverse effects or discomfort experienced by participants during their interaction with the virtual environment. It encompasses 16 items categorized into three subscales: oculomotor, disorientation, and nausea. Each item is rated on a scale from 0 to 3, and the overall score ranges from 0 to 48. Higher scores indicate higher discomfort
Technology Acceptance | The initial, second, fifth, ninth, thirteenth, and final intervention sessions.
  The questionnaire assesses an individual's confidence and attitude levels toward technology. Seven sub-scales will be used, including Perceived Ease of Use (4 items), Perceptions of External Control (4 items), Computer Anxiety (4 items), Perceived Enjoyment (3 items), Output Quality (3 items), Result Demonstrability (4 items), and Behavioral Intention (3 items). It employs a seven-point Likert scale, the score ranges from 25 to 175. Higher scores indicate a higher technology acceptance.

REFERENCES:
- [Derived] Chen IC, Wu CY, Hu YL, Huang YM. Development and Validation of Virtual Reality Cognitive Training for Older Adults with Mild Cognitive Impairment: Protocol for a Mixed-Methods Program Evaluation Study. Clin Interv Aging. 2024 Nov 9;19:1855-1865. doi: 10.2147/CIA.S471547. eCollection 2024. PMID 39539569